CLINICAL TRIAL: NCT00592332
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Question 2
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Q2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steve Davis, Department Chair, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: IRB#040908-HAAF-T1DM-Q2; DK69803
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Alprazolam; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Hyperinsulinemic glucose clamp with Xanax given orally at beginning of each 2 hour clamp on day 1.
  Interventions: Drug: Alprazolam
- 1 (Experimental): Hyperinsulinemic glucose clamp in group with no drug.
  Interventions: Other: control group

INTERVENTIONS:
Drug: Alprazolam — 1 mg alprazolam given orally 60 minutes prior to each 2 hour glucose clamp on day 1 (x2)
  Other Names: Xanax
  Arms: 2
Other: control group — control group is two hyperinsulinemic glucose clamps on day 1 with no drug given.
  Arms: 1

SUMMARY:
Alprazolam (Xanax) will blunt the body's ability to defend itself from low blood sugar.

DETAILED DESCRIPTION:
Due to the fundamental importance of glucose as a cerebral fuel, a complex and redundant counterregulatory response to hypoglycemia exists in man. Some studies have shown that prior activation of GABA(A) receptors may result in blunting of counterregulatory responses during next day hypoglycemia.

The Specific Aim is to determine if repeated activation of GABA(A) receptors using Alprazolam will result in blunting of neuroendocrine, ANS and metabolic counterregulatory mechanisms during next day hypoglycemia in T1DM and healthy man.

ELIGIBILITY:
Inclusion Criteria:

* 16 (8 males, 8 females) Type 1 diabetes patients aged 18-45 yr.
* 16 (8 males, 8 females) healthy controls aged 18-45 yr.
* HbA1c > 7.0% (Type 1 diabetes patients)
* Had diabetes for 2-15 years (Type 1 diabetes patients)
* No clinical evidence of diabetic tissue complications (Type 1 diabetes patients)
* Body mass index 21-30 kg · m-2
* Normal bedside autonomic function
* Normal results of routine blood test to screen for hepatic, renal, and hematological abnormalities
* Female volunteers of childbearing potential: negative HCG pregnancy test

Exclusion Criteria:

* Prior history of poor health: any current or prior disease condition that alters carbohydrate metabolism and prior cardiac events and/or evidence for cardiac disease
* Hemoglobin of less than 12 g/dl
* Abnormal results following screening tests
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with known liver or kidney disease
* Subjects taking steroids
* Subjects taking beta blockers
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Catecholamine levels | Comparative study performed every 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States